CLINICAL TRIAL: NCT01571661
Title: A Double Blind, Randomized, Placebo Controlled, Single-dose Escalation, First-time-in-human Crossover Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Ascending Doses of GSK189075A in Healthy Subjects and in Subjects With Type 2 Diabetes Mellitus
Brief Title: A First-time-in-human Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Ascending Doses of GSK189075A in Healthy Subjects and in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: KG219017
Record Dates: First submitted 2012-03-15; First posted 2012-04-05 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: KGT-1142; safety; pharmacokinetics; single-dose escalation; tolerability
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Part A Treatment 1 (Experimental): GSK189075A 20mg
  Interventions: Drug: GSK189075A
- Part A Treatment 2 (Experimental): GSK189075A 50mg
  Interventions: Drug: GSK189075A
- Part A Treatment 3 (Experimental): GSK189075A 150mg
  Interventions: Drug: GSK189075A
- Part A Treatment 4 (Experimental): GSK189075A 500mg
  Interventions: Drug: GSK189075A
- Part A Treatment 5 (Experimental): GSK189075A 1000mg
  Interventions: Drug: GSK189075A
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- Part B Low dose (Experimental): low dose chosen from Part A
  Interventions: Drug: GSK189075A
- Part B High Dose (Experimental): high dose chosen from Part A
  Interventions: Drug: GSK189075A

INTERVENTIONS:
Drug: GSK189075A — 20mg, 50mg, 150mg, 500mg, 1000mg or Placebo
  Arms: Part A Treatment 1; Part A Treatment 2; Part A Treatment 3; Part A Treatment 4; Part A Treatment 5; Part B High Dose; Part B Low dose
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a double blind, randomised, placebo controlled, single dose escalation, first-time-in-human, 5-way crossover study to assess the safety, tolerability, pharmacokinetic and pharmacodynamic parameters of ascending doses of GSK189075A in healthy subjects (Part A). Single doses will be given to 10 healthy subjects. The planned doses are 20mg, 50mg, 150mg, 500mg, and 1000mg. Each subject will receive 4 of the 5 active doses and a placebo separated by a washout of 5-10 days. A second cohort of 6 subjects with type 2 diabetes mellitus will receive 2 active doses and a placebo along with oral glucose in a three-way, randomised, placebo controlled, crossover design to assess glucose lowering following GSK189075A administration (Part B). Blood samples will be taken throughout the study day for pharmacokinetic analysis of prodrug and metabolites. Safety will be assessed by measurement of blood glucose, blood pressure, heart rate, ECGs, laboratory safety screens, and collection of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Women must be of non-childbearing potential. Non-childbearing potential is defined as: Post-menopausal females defined as being amenorrhoeic for greater than one year with an appropriate clinical profile, e.g., age appropriate, history of vasomotor symptoms. However, if indicated, this should be confirmed by estradiol and FSH levels consistent with menopause (according to local laboratory ranges) Pre-menopausal females with a documented (medical report verification) hysterectomy or tubal ligation.
* A negative pre-study urine drug screen. A minimum list of drugs that will be screened includes amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* Negative results for hepatitis C antibodies, hepatitis B surface antigen and HIV at screening, or have documented negative test results within the last 6 months.
* Signed and dated written informed consent prior to admission to the study.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.
* Subjects with the following clinical laboratory values: ALT and AST < 2 times the upper limit of normal at screening and prior to the first dose; fasting triglycerides < 400mg/dL at screening and prior to first dose; bilirubin < 1.5 times the upper limit of normal at screening and prior to the first dose (total; subjects above this limit may only be included if direct bilirubin is within normal limits).

Other values must be within the normal range or not clinically significant at screening and check-in. Abnormal values, deemed clinically significant by the principal investigator, must be cleared by the medical monitor at GSK.

* Additional inclusion criteria for subjects in Part A: A subject will be eligible for inclusion in Part A of this study only if all of the following criteria apply: Healthy adult subjects aged 18 to 55 years inclusive, male and female subjects of non-childbearing potential.
* Body weight greater than or equal to 50kg for men and greater than or equal to 45kg for women and BMI within the range 19.0 to 30.0kg/m2 inclusive.
* Healthy as judged by responsible physician. No clinically significant abnormality identified on the medical or laboratory evaluation, including 12-lead ECG. A subject with a clinically significant abnormality, or laboratory parameters outside the reference range for this age group may be included only if the Investigator and Sponsor's Medical Monitor considers that the finding will not introduce additional risk factors and will not interfere with the study procedures.
* Part B: A subject will be eligible for inclusion in Part B of this study only if all of the following criteria are met: Subjects with documented type 2 diabetes mellitus diagnosis (diagnosed not less than 6 months; HbA1c less than or equal to 10 % and FPG < 280 mg/dL at screening) who are either controlled by diet alone or monotherapy for a minimum of 3 months with either oral sulfonylureas, rosiglitazone, metformin, or acarbose. They must be willing/able to discontinue these medications during each dosing occasion for up to 72 hours (from check-in into the research unit until released after the last study assessment for each dosing period).
* Adult men and women between 30 - 60 years inclusive. Women must be of non-childbearing potential.
* BMI within the range 22 35kg/m2 inclusive.
* Subjects taking stable regimens of medications commonly used as prevention in diabetics (aspirin, ACE inhibitors, and statins) will be allowed if their dose regimen(s) remain constant throughout the study period. Concurrent usage of prescribed medications other than the medications listed above may be allowed to continue only with Sponsor's consent.
* No significant concomitant health problems other than type 2 diabetes mellitus and otherwise healthy as judged by a responsible physician.
* Systolic/Diastolic blood pressure: greater than or equal to 80/60 mmHg and less than or equal to 150/95 mmHg at screening.

Exclusion Criteria:

* History or presence of allergy to the study drug or drugs of this class or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* History or presence of gastrointestinal, hepatic or renal disease, or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs. Any acute gastrointestinal illness within 2 weeks prior to dosing.
* Use of diuretics, systemic corticosteroids, or any other medication that may result in electrolyte depletion, within 3 weeks of any scheduled dose.
* Blood electrolyte (K, Na, Cl, Mg or Ca or bicarbonate) values outside of the reference range at screening and admission. No deviation will be permitted unless there has been discussion on an individual basis between sponsor and investigator for the following parameters: sodium, potassium, chloride, bicarbonate, calcium and magnesium.
* If participation in the study will result in the subject having donated more than 1,500mL blood (males) or 1,000mL (females) in the previous 12 months and 6. where participation in study would result in donation of blood in excess of 550mL within a 56-day period.
* As a result of the medical interview, physical examination for screening investigations, the Physician Responsible considers the volunteer unfit for the study.
* They have suffered a urinary tract or bladder infection within 4 weeks of the start of the study.
* Abuse of alcohol
* Significant renal disease
* Any clinically significant abnormality identified on the medical or laboratory evaluation, including 12-lead ECG and 24 h Holter monitoring. A subject with a clinically significant abnormality or laboratory parameters outside the reference range for this age group may be included only if the Investigator and Sponsor's Medical Monitor consider that the finding will not introduce additional risk factors and will not interfere with the study procedures
* Participation in a study trial with any drug of new chemical entity within 90 days prior to the start of the study.
* Male subject unwilling to abstain from, or use a condom during sexual intercourse with a pregnant or lactating female; or male subject unwilling to use a condom plus another form of contraception (e.g., spermicide, IUD, birth control pills taken by female partner, diaphragm with spermicide) during sexual intercourse with a female who could become pregnant. Any male subject unwilling to adhere to the above contraceptive criteria from administration of study medication until completion of follow-up procedures.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication and until released after the last study assessment after the last dosing period, unless in the opinion of the Investigator and Sponsor the medication will not interfere with the study procedures or compromise subject safety.
* Part A: A subject will not be eligible for inclusion in Part A of this study if the following applies: Past or present disease, which as judged by the Investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease and endocrine disease.
* Part B: A subject will not be eligible for inclusion in Part A of this study if any of the following criteria apply: Currently requiring insulin therapy, or has been on insulin therapy for the previous 3 months prior to the screening examination.
* Medically unable or unwilling to discontinue their oral antidiabetic medications for up to 72 hours (from check-in into the research unit until released after the last study assessment for each dosing period).
* Past or present disease (other than type 2 diabetes mellitus) as judged by the Investigator, which may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease and endocrine disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2004-09; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability change from baseline in laboratory assessments | Part A: Approximately 58 days and Part B: Approximately 38 days.
  Hematology, Clinical Chemistry, Urinalysis
Safety and tolerability change from baseline in electrocardiaogram (ECG) reading | Part A: Approximately 58 days and Part B: Approximately 38 days.
  12-lead ECG and continuous ECG monitoring.
Safety and tolerability change from baseline in fluid intake | FPart A: Approximately 58 days and Part B: Approximately 38 days.
  urine output, and the number of micturations will be recorded.
Safety and tolerability change from baseline in electrolytes | Part A: Approximately 58 days and Part B: Approximately 38 days.
  Blood electrolyte concentrations (Na, K, Cl, Ca, Mg and bicarbonate)
Safety and Tolerability change from baseline in creatinine clearance | Part A: Approximately 58 days and Part B: Approximately 38 days.
  creatinine clearance (24-hours [h])
Composite of pharmacokinetic parameters of GSK189075A, GSK189074A, and GSK279782A | Part A: up to 24 hours post dose for five periods. Part B: For 24 hours post dose for 3 periods. Collected at the following: pre-dose, and 10 min, 20 min, 30 min, 45 min, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, , 8, 12, 16 and 24h post-dose.
  Area under the plasma concentration-time curve [AUC(0 last)], Area under the plasma concentration-time curve [AUC(0-infinity)], Maximum observed plasma concentration (Cmax), Time to maximum observed plasma concentration (tmax), Plasma elimination half-life (t1/2), Area under the plasma concentration-time curve for the metabolite [AUCm(0-last)]/ Area under the plasma concentration-time curve for the parent [AUCp(0-last)], and AUCm(0-infinity)/AUCp(0-infinity) ratios.
Parts A and B: plasma glucose concentrations in healthy subjects | Part A: up to 24 hours post dose for five periods. Part B: For 24 hours post dose for 3 periods.
Parts A and B: Urine chemistry lab measurements | measurements will be obtained pre-dose, and over the following intervals: 0-2, 2-4, 4-6, 6-8, 8-12, and 12-24h during the dosing period.
  Urine samples for creatinine, glucose, and electrolytes (Na, K, Cl) measurements will be obtained.
Part B: Plasma glucose and insulin concentrations concentrations in subjects with type 2 diabetes mellitus following a 50g oral glucose challenge. | On day -2 predose and at 0.5, 1, 1.5, 2, 4, 4.5, 5, 6, 8, 10, 12 and 24h.
Safety and Tolerability as assessed by numbers of adverse events | Part A: Approximately 58 days and Part B: Approximately 38 days.
  number of adverse events collected during study
Safety and Tolerability as assessed by change from baseline in vital sign measurements | Part A: Approximately 58 days and Part B: Approximately 38 days.
  Blood pressure and heart rate.
urine glucose concentrations in subjects with type 2 diabetes mellitus following a 50g oral glucose challenge. | On day -2 predose and at 0.5, 1, 1.5, 2, 4, 4.5, 5, 6, 8, 10, 12 and 24h.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Kapur A, O'Connor-Semmes R, Hussey EK, Dobbins RL, Tao W, Hompesch M, Smith GA, Polli JW, James CD Jr, Mikoshiba I, Nunez DJ. First human dose-escalation study with remogliflozin etabonate, a selective inhibitor of the sodium-glucose transporter 2 (SGLT2), in healthy subjects and in subjects with type 2 diabetes mellitus. BMC Pharmacol Toxicol. 2013 May 13;14:26. doi: 10.1186/2050-6511-14-26. PMID 23668634